CLINICAL TRIAL: NCT06050707
Title: MR-Adaptive Radiation Therapy for Anal Cancer With EScalated-Treatment in a Risk-Optimized Approach
Acronym: MAESTRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5323
Record Dates: First submitted 2023-08-18; First posted 2023-09-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Anal Squamous Cell Carcinoma
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy - Low risk group — 20 fractions completed in 4 weeks
Radiation: Radiotherapy - Standard risk group — 25 fractions completed in 5 weeks
Radiation: Radiotherapy - Intermediate risk group — 30 fractions completed in 6 weeks
Radiation: Radiotherapy - High risk group — 35 fractions completed in 7 weeks

SUMMARY:
The proposed study is a phase II, single arm, open-label trial of MR-guided radiation therapy (RT) with risk stratified RT dose selection in patients with anal cancer. Based on previous data, a risk adaptive treatment approached is proposed in 4 groups: Low risk, standard risk, intermediate risk, and high risk. Human papillomavirus (HPV) DNA will be analyzed to identify novel biomarkers that predict chemoradiotherapy (CRT) response and toxicity.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a risk-stratified dose of treatment (radiation dose and chemotherapy number of cycles) based on predefined clinical and biological biomarkers for anal squamous cell carcinoma (SCC). Radiotherapy will be delivered on the MR-Linac for image-guided-radiation therapy (IGRT). Patients will be followed for up to 5 years after radiotherapy and be required to complete questionnaires and clinic visits. Patients have the option to complete blood and tissue samples during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven diagnosis of anal SCC. This may include tumors of non-keratinizing histology such as basoloid or cloacogenic histology. Individuals with squamous cell carcinoma of the anal margin are eligible.
* Clinical stage T1-4 N0-1 M0 (the Union for International Cancer Control (UICC) / the American Joint Committee on Cancer (AJCC) 8th Ed)
* Patients must be eligible for definitive RT or CRT
* Must be ≥ 18 years of age
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Previous chemotherapy, RT or curative-intent surgical treatment (i.e. APR) for anal cancer.
* Any previous RT to the abdomino-pelvic region that would result in overlap of RT volume for the current study.
* Individuals with a history of a different malignancy except if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in locoregional failure (LRF) at Year 2 | 2 years
  Any local or regional failure from the date of registration to the date of any of the local or regional failure.

SECONDARY OUTCOMES:
Presence of distant metastasis (DM) | 5 years
  Clear clinical/radiographic evidence of distant metastases in the lung, bone, brain, liver or other distant sites.
Colostomy rate | 5 years
  The presence of a colostomy until colostomy removal.
Disease free survival (DFS) | 5 years
  The time from the date of registration to the date of first record of any of the following events including local, regional, distant failure, or death due to any cause.
Overall survival (OS) | 5 years
  The time from the date of registration to the date of death for any cause.
Physician-reported toxicities | 5 years
  Using the National Cancer Institute (NCI) Common Terminology Criteria of Adverse Events (CTCAE) V.5.
Patient Reported Outcomes | 5 years
  Using the Common Terminology Criteria of Adverse Events
Quality of life (QOL) | 5 years
  Based on the completion of the European Organisation For Research And Treatment Of Cancer (EORTC-C30) questionnaire. The EORTC-C30 questionnaire is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients.
Quality of life (QOL) | 5 years
  Based on the completion of the European Organisation For Research And Treatment Of Cancer (EORTC-AN27) questionnaire. EORTC QLQ-ANL27 includes four quality of life domains: pain, bowel, sexual and stoma care problems and five single item (frequent urination, keeping clean, proximity to toilet, lower limb oedema, planning activities)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Austin Health, Heidelberg, Victoria, Australia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No